CLINICAL TRIAL: NCT02292277
Title: Evaluation of Ticagrelor Pharmacokinetics in Patients With Non-ST Elevation Myocardial Infarction After a 180 mg Ticagrelor Loading Dose
Brief Title: Ticagrelor Pharmacokinetics in NSTEMI
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Jan van der Linden, Professor, Karolinska University Hospital
Other Study IDs: 2014/1174-31/1
Record Dates: First submitted 2014-11-05; First posted 2014-11-17 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Myocardial Infarction
Keywords: Ticagrelor; Pharmacokinetics; Platelet Aggregation; Platelet Function Tests
MeSH Terms: conditions — Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of venous blood will be collected into lithium-heparin tubes, centrifuged at 1500 g at 4ºC for 10 min within 30 min of blood sampling at the following time points: pre-dose, 1, 2, 3, 4, 5, and 6 hours post-dose, as shown in the table below. For P2Y12-antagonist naïve patients and controls, sampling of venous blood into Hirudin tubes for pharmacodynamics evaluation will be performed for analysis using an ADP-induced platelet aggregation assay.
  The resulting plasma samples will then be stored below minus 20ºC until analyzed. Plasma concentrations of ticagrelor and its active metabolite AR-C124910XX will be determined by validated methods (high-performance liquid chromatography and tandem mass spectrometry detection; LC-MS/MS) at a certified laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NSTEMI patients: Subjects eligible for the study will be ticagrelor naïve patients with NSTEMI presenting at the emergency room. Upon arrival to the emergency room written informed consent will be obtained before the patients receive their 180 mg loading dose of ticagrelor, as prescribed by the responsible physician.
  Interventions: Drug: Ticagrelor
- SCAD controls: Patients with stable coronary artery disease (SCAD) planned for elective angiography. If PCI is to be performed and if the responsible physician decides to administrate a loading dose of 180 mg ticagrelor, written informed consent will be obtained before loading dose and blood sampling.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Oral loading dose of 180 mg ticagrelor.
  Other Names: Brilique

SUMMARY:
Patients with myocardial infarction, which does not include all layers of the heart's muscle wall are common and they often receive pharmacological treatment with the platelet inhibiting drug ticagrelor. However, the drug uptake after an oral dose of 180mg ticagrelor has not been thoroughly studied in these patients.

The present study will evaluate ticagrelor uptake and platelet aggregation after a 180 mg loading dose ticagrelor in these patients.

DETAILED DESCRIPTION:
This study is to be considered as an observational prospective case-controlled study, according to the Swedish Medical Product Agency (MPA), in response to our enquiry. This is due to lack of intervention in routine medical treatment.

Patients with non-ST elevation myocardial infarction (NSTEMI) are common, but the pharmacokinetic properties of ticagrelor in the acute phase have, to the best of our knowledge, not been thoroughly studied in these patients.

The present study will evaluate ticagrelor uptake and platelet aggregation after a 180 mg loading dose ticagrelor in NSTEMI patients and compare results with a control group of patients with stable coronary artery disease.

Hypotheses/questions The stress reaction from suffering an NSTEMI causes delayed absorption and possibly delayed and lowered maximal plasma concentrations after a loading dose ticagrelor and thus a delayed and possibly impaired inhibition of platelet aggregation.

Method Study population Subjects eligible for the study will be ticagrelor naïve patients with NSTEMI presenting at the emergency room at Södersjukhuset. Upon arrival to the emergency room written informed consent will be obtained before the patients receive their 180 mg loading dose of ticagrelor if the responsible physician choses this therapy. Inclusion criteria: 1) a diagnosis of NSTEMI (i.e relevant symptoms associated with ischemic ECG changes (not categorized as STEMI) and/or relevantly increased cardiac markers); 2) an indication for a 180 mg ticagrelor loading dose.

Control group Patients with stable coronary artery disease presenting at the cardiology clinic at Södersjukhuset. A single 180 mg loading dose of ticagrelor will be administrated if the responsible physician choses this therapy. Inclusion criteria. The inclusion criterion for the control group will be documented stable coronary artery disease. Exclusion criteria: 1) ACS within the last 3 months; 2) Age <18 years; 3)Administration of ticagrelor during the week before inclusion; 4) Treatment with glycoprotein IIb/IIIa antagonists within 48 hours before inclusion; 5) Ongoing morphine treatment.

Study procedures and methods Samples of venous blood will be collected into lithium-heparin tubes, centrifuged at 1500 g at 4ºC for 10 min within 30 min of blood sampling at the following time points: pre-dose, 1, 2, 3, 4, 5, and 6 hours post-dose, as shown in the table below. For P2Y12-antagonist naïve patients and controls, sampling of venous blood into Hirudin tubes for pharmacodynamics evaluation will be performed for analysis using an ADP-induced platelet aggregation assay (Multiplate®, Roche Diagnostics International Ltd, Rotkreuz, Switzerland).

The resulting plasma samples will then be stored below minus 20ºC until analyzed. Plasma concentrations of ticagrelor and its active metabolite AR-C124910XX will be determined by validated methods (high-performance liquid chromatography and tandem mass spectrometry detection; LC-MS/MS) at a certified laboratory (Covance Laboratories Inc.).

Statistical analysis The median Tmax in the control group with stable coronary artery disease can be expected at approximately 2 hours after a 180 mg loading dose. The range of the Tmax in patients with stable coronary artery disease receiving a 180mg loading dose was between 1 and 8 hours. A rough standard deviation estimate of 1.25 hours was obtained from this range using the formula (ln (maxT⁡max) - ln (minTmax))/k from a statistical textbook by Dixon et al. A statistician estimated k to 9.5 from a natural distribution table. The estimated standard deviation of 0.22 on the logarithm scale was then calculated using the calculation above. For the study group with NSTEMI, a larger standard deviation can be expected and was estimated with the following formula provided by the statistician: sqrt((0.22^2 )× 2)) =0.31.

To make a sample size calculation possible, the above calculated standard deviations were anti-logged using the exponential function and found to be 1.25 hours and 1.36 hours, respectively.

For the power calculation, a 50% delay in median ticagrelor Tmax (1 hour delay) was considered, as this can be regarded as a clinical significant difference. A power calculation with the above described time to Tmax and estimated standard deviations, showed that a study with 80% power would require 40 patients in the study group and 20 patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of NSTEMI (i.e relevant symptoms associated with ischemic ECG changes (not categorized as STEMI) and/or relevantly increased cardiac markers);
* An indication for a 180 mg ticagrelor loading dose.

Exclusion Criteria:

* Ticagrelor contraindication, including

  * Hypersensitivity to the active substance or to any of the excipients listed in section 6.1
  * Active pathological bleeding
  * History of intracranial haemorrhage
  * Moderate to severe hepatic impairment.
  * Co-administration of ticagrelor with strong CYP3A4 inhibitors (e.g., ketoconazole,clarithromycin, nefazodone, ritonavir, and atazanavir) is contraindicated, as co-administration may lead to a substantial increase in exposure to ticagrelor
* Age <18 years
* Administration of ticagrelor during the week before inclusion
* Treatment with glycoprotein IIb/IIIa antagonists within 48 hours before inclusion
* Ongoing morphine treatment. However, if patients with NSTEMI without morphine treatment are rare, this exclusion criterion of the protocol may have to be re-evaluated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at emergency department and angiography laboratory
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Tmax ticagrelor | Within 6 hours after oral intake
  Time to maximum concentration (Tmax) of ticagrelor after a 180 mg loading dose.

SECONDARY OUTCOMES:
Tmax AR-C124910XX | Within 6 hours after oral intake
  Tmax of the active ticagrelor metabolite AR-C124910XX
Pharmacodynamic response | Predose, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours post dose.
  Evaluation of relationship between plasma concentrations of ticagrelor and platelet aggregation (Aggregation Units) response in P2Y12-antagonist naïve subjects after a 180 mg ticagrelor loading dose
HPR at 2 hours | 2 hours after oral intake
  Frequency of high-on-treatment platelet reactivity (HPR) 2 hours after a 180 mg ticagrelor loading dose

CONTACTS AND LOCATIONS:
Overall Officials: Jan van der Linden, MD, PhD, Principal Investigator — Dept of Molecular Medicine and Surgery, Karolinska Institutet
Locations (1):
- Södersjukhuset, Stockholm, Sweden